CLINICAL TRIAL: NCT04935268
Title: Demographic Differences in Patients With Abdominal Aortic Aneurysm and Surgical Features of Treatment
Status: Completed | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Ryazan Medical University
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-08

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study of demographics and risk factors for abdominal aortic aneurysms, allows to individualize treatment approaches.

Determining of the results of treatment of patients who requires a late open conversion after EVAR will allow to develop the surgical approach and the selection of the optimal type of surgical treatment.

Determination of genetic polymorphisms will reduce the number of postoperative complications by predicting of possible complications in the long term period.

ELIGIBILITY:
Inclusion Criteria:

* Infrarenal Aortic Aneurysm

Exclusion Criteria:

* Other Aneurysms

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients wit infrarenal Aortic Aneurysms
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Survival | 1-60 Month
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Igor A Suchkov, Prof, Study Director — Ryazan State Medical University; Egan Kalmykov, Dr, Principal Investigator — Clinic of Vascular Surgery, Frechen
Locations (1):
- Egan Kalmykov, Frechen, Please Select, Germany

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: SAP, CSR